CLINICAL TRIAL: NCT01521520
Title: Ferumoxytol Enhanced Magnetic Resonance Imaging of Type 1 Diabetes Progression
Brief Title: Imaging of Type 1 Diabetes Progression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jason Gaglia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor-Investigator, Jason Gaglia, Research Scientist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 2011P001957; P01AI054904 (NIH)
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; magnetic resonance imaging; insulitis; ferumoxytol
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Clinical Type 1 Diabetes: This group will be subdivided into individuals with recent onset clinical type 1 diabetes (within 6 months of diagnosis), latent autoimmune diabetes of the adult, and longer standing type 1 diabetes.
  Interventions: Drug: ferumoxytol
- High Risk Pre-Type 1 Diabetes: High risk pre-type 1 diabetes is defined as first degree family relative with type 1 diabetes and at least one islet autoantibody marker (GAD, IAA, or IA-2).
  Interventions: Drug: ferumoxytol
- Low Risk Pre-Type 1 Diabetes: Low risk pre-type 1 diabetes is defined as first degree family relative with type 1 diabetes but no islet autoantibody markers (GAD, IAA, or IA-2).
  Interventions: Drug: ferumoxytol
- Normal Control: Normal control is based on history with no known history or family history of type 1 diabetes.
  Interventions: Drug: ferumoxytol

INTERVENTIONS:
Drug: ferumoxytol — Ferumoxytol at a dose of between 1 and 6 mg iron/kg body weight (maximum 510 mg/injection) will be administered via intravenous injection. Ferumoxytol will be administered with each series of MRIs.
  Other Names: Feraheme

SUMMARY:
Type 1 diabetes results from the autoimmune destruction of the insulin-producing beta cells of the islets of Langerhans of the pancreas. Initially, diabetes is usually clinically silent with immune cells invading the pancreatic islets, a process termed insulitis, which eventually leads to loss of beta cells in the islets. If enough beta cells are destroyed, the body can not make enough insulin to maintain blood sugars in the normal range and clinical diabetes develops. The purpose of this study is to assess the ability of magnetic resonance imaging with ferumoxytol to detect changes in the pancreas associated with the insulitis of type 1 diabetes.

DETAILED DESCRIPTION:
This study is designed to monitor changes associated with the development of autoimmune diabetes. A magnetic resonance imaging (MRI) based technique will be used to noninvasively measure changes within the pancreas associated with the development of autoimmune diabetes. The iron-containing drug ferumoxytol will be used as an intravenous MRI contrast agent for this study.

Individuals will be asked to participate one time, for 1-year, or over a 2-year period. During the development phase of the study, each imaging series will consist of 3 or more MRI scans. At the initial imaging visit a pre-ferumoxytol scan will be done, followed by ferumoxytol injection, and then an immediate post-injection scan. The subsequent scans will be concluded within 96 hours of ferumoxytol injection (typically at 48 hours). Those who participate for 1-year will have repeat imaging at approximate times 0, 6 months, and 12 months. Those who participate for 2-years will have repeat imaging at approximate times 0, 3, 6, 12, 18, and 24 months after enrollment.

Measurements of autoimmunity and metabolic parameters (collected as part of collaborating diabetes clinical studies) will be used in the data analysis for the longitudinal portion of the study. Stimulated C-peptide will be measured as a marker of endogenous insulin production capacity and beta-cell mass.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a collaborating diabetes clinical trial
* Able to understand written consent document and HIPAA authorization prior to initiation of study related procedures and are willing to participate

Exclusion Criteria:

* Known allergy to ferumoxytol or iron
* Individuals who are pregnant or lactating
* Iron saturation above the upper limit of normal
* Individuals with a counter-indication to MRI, such as the presence of metallic prostheses or implanted metal device (e.g., infusion pump, defibrillator)
* Individuals with known clinical conditions that may lead to iron overload including hemochromatosis, cirrhosis, or sickle cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from those already participating in diabetes clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2012-01

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gaglia, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gaglia JL, Guimaraes AR, Harisinghani M, Turvey SE, Jackson R, Benoist C, Mathis D, Weissleder R. Noninvasive imaging of pancreatic islet inflammation in type 1A diabetes patients. J Clin Invest. 2011 Jan;121(1):442-5. doi: 10.1172/JCI44339. Epub 2010 Dec 1. PMID 21123946